CLINICAL TRIAL: NCT00211926
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate Safety and Immunogenicity of StaphVAX®, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine, in Adult Patients Receiving an Orthopaedic Prosthetic Implant
Brief Title: StaphVAX Immunogenicity in Orthopedic Implant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Matt Hohenboken, MD, PhD/ Executive Director Clinical and Medical Affairs, Nabi Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nabi-1365
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Staphylococcal Infections; Joint Prosthesis
Keywords: vaccine; Staphylococcus aureus vaccine
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- StaphVAX (Experimental)
  Interventions: Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Conjugate
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Conjugate — single dose of vaccine containing 100 mcg of each serotype conjugate
  Arms: StaphVAX
Biological: placebo — single dose of placebo
  Arms: Placebo

SUMMARY:
S. aureus is the most common pathogen involved in prosthetic joint infection. StaphVAX® is a vaccine to prevent these infections, which conjugates the purified capsular polysaccharides of S. aureus to a carrier protein. It is currently being evaluated for future licensing. This study aims to demonstrate the safety and immunogenicity of a single dose of StaphVAX in patients who are candidates for knee or hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* candidate for knee or hip replacement
* expectation of protocol compliance
* negative pregnancy test, where appropriate

Exclusion Criteria:

* known S. aureus infection in the prior 3 months
* infection in the prior 2 weeks
* Known HIV infection
* immunomodulatory drugs
* Malignancy (other than basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or early stage prostate cancer)
* Hypersensitivity to components of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
serotype-specific antibody concentrations | 6 weeks after dose

SECONDARY OUTCOMES:
serotype-specific antibody concentrations | several other time points after dose, up to 365 days
safety: adverse events | 0-365 days

CONTACTS AND LOCATIONS:
Overall Officials: Preston Holley, MD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- Cllinical Research Asociates of Tidewater, Norfolk, Virginia, United States